CLINICAL TRIAL: NCT04921150
Title: Standardized Management of Complex Twins
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Caixia Liu (Other)
Collaborators: Shengjing Hospital (Other)
Responsible Party: Sponsor-Investigator, Caixia Liu, Clinical Professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SMOCT
Record Dates: First submitted 2021-05-26; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Twins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: standardization management — Apply standardization management to improve the outcomes of pregnancy

SUMMARY:
At present, the incidence of monochorionic twins in all pregnancies is around 3-5‰ worldwide.In 2019, the twin Committee of China Maternal and Child Health Association conducted statistics from 48 medical units all over the country, showing that there were 4,876 cases of monochorionic twins, accounting for 10.2‰ of all pregnancies.In addition to increased incidence of preterm delivery, miscarriage, and maternal complication, the unique placental vascular structure of monochorionic twins is associated with complex fetal complication such as twin-twin transfusion syndrome, selective intraurine growth restriction, twin anaemia-erythrocytosis sequence, twin reversed arterial perfusion sequence, one of twin with dysplasia, twins with single amniotic sac and conjunctions are common. At present, there is no unified standard for the diagnosis and treatment of these complicated twins, and various treatment methods have a great impact on the pregnancy outcome and fetal prognosis.Therefore, the standardized management of complex twins benefits diagnosis and treatment of complex twins and improves fetal prognosis.

ELIGIBILITY:
Inclusion Criteria:

complex twin disease 18-45 years

Exclusion Criteria:

single pregnancy normal twin pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Standardized management system of twin pregnancy clinic | 1 year
  S/D score and Apgar score of complex twin pregnancy assessed by clinical doctors

IPD SHARING:
Plan to Share IPD: No